CLINICAL TRIAL: NCT04637711
Title: Randomized Controlled Trial for 'Focus Clearing + Whole Breast Exploration and Washing + One-Stage Micro Plastic Surgery' Treatment for Granulomatous Lobular Mastitis
Brief Title: Surgical Intervention for Refractory Granulomatous Lobular Mastitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Ph D, MD, Chair, Department of Thyroid and Breast Surgery, Zhongnan Hospital of Wuhan University, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYL[2020091]
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Refractory Granulomatous Lobular Mastitis
Keywords: granulomatous lobular mastitis ；refractory；surgery
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific surgical Intervention (Experimental): Focus clearing + whole breast exploration and washing + one-stage micro plastic surgery
  Interventions: Procedure: Focus clearing + whole breast exploration and washing + one-stage micro plastic surgery No Intervention: Extensive lesion excision
- Extensive lesion excision (No Intervention)

INTERVENTIONS:
Procedure: Focus clearing + whole breast exploration and washing + one-stage micro plastic surgery No Intervention: Extensive lesion excision — Only visible lesions and necrotic tissues, such as abscess cavity, sinus tract and fistula, were removed intraoperatively, while normal glands and fat were retained. Preoperative ultrasound was used to locate the lesion area and then the surgical incision was designed. Intraoperative ultrasound examination of latent small lesions, resection of lesions visible under ultrasound, and then a full breast exploration, one finger page incision interval.Radially cut from the base to the subcutaneous, lesions were found and treated locally. After removal of lesion, fully using the syringe, in turn, use of 3% hydrogen peroxide solution, 1% eniodine, saline water is widely jet pulse washing, and around the lesions base. After rinsing, soak in 1% active iodine for 10min, then rinse with normal saline until the liquid is clear. Breast tumor Surgery (Oncoplastic Breast Surgery, OBS) core technology (volume replacement and volume replacement).
  Arms: Specific surgical Intervention

SUMMARY:
Granulomatous lobular mastitis (GLM) belongs to a group of benign diseases, which is mainly treated with glucocorticoids and surgical treatment. Nowadays, in China, surgical treatment has gradually become the mainstream, but the timing and the extent of surgery are still controversial, and different literatures report that the recurrence rate after surgery is 20-50%. Empirical lesion resection is generally used. We believe that the main reason for the high recurrence rate is the incomplete removal of the breast lesions. Because GLM is often characterized with microabscesses formation, empirical resection is likely to have residual lesions that are not visible to the naked eye. In order to reduce the postoperative recurrence rate and protect the breast appearance as much as possible, we propose a surgical plan : granulomatous lobular mastitis "lesion removal + whole breast exploration and flushing + one-stage microplastic surgery". The purpose of this study was to compare this surgical scheme of granulomatous lobular mastitis with existing surgical schemes, and to compare the overall benefits of the two for patients with GLM. We aim to protect the breast appearance on the premise of low recurrence, improve the quality of life of GLM patients, and standardize GLM surgical schemes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with granulomatous lobular mastitis
* Patients without surgical treatment;
* Extensive lesions involving two or more quadrants of the breast, or accompanied by abscess, sinus fistula formation, skin rupture and other complex lesions;
* Patients volunteered to participate in the study after informed consent.

Exclusion Criteria:

* Patients were diagnosed with mastitis with other definite etiology confirmed by pathology
* Patients who chose conservative treatment and did not receive surgical treatment
* Combined with other basic diseases, unable to tolerate surgery
* Patients in pregnancy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | Up to 2 years
  Inflammatory changes, mass, abscess or fistula formation, nodular erythema of the upper and lower extremities and joint pain occurred in the ipilateral breast within one year after surgery was defined as recurrence.

SECONDARY OUTCOMES:
Breast appearance and cosmetic effect score | Up to 2 years
  Refer to Harris standard to evaluate postoperative cosmetic effect. Specify the breast appearance and cosmetic effect rating table.
Surgical incision healing time | Up to 2 months
  Surgical incision healing time was defined as the time from the first day after the operation to the healing time of the surgical incision. The wound surface was dry, there was no effusion, and no surgical incision complications occurred

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No